CLINICAL TRIAL: NCT02906150
Title: Thymosin Alpha 1 Plus Maintenance Therapy With the Standard of Care (SoC) Chemotherapy Plus Cisplatin (or Carboplatin) in Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC), EGFR Wild Type
Brief Title: Thymosin Alpha 1 Plus Maintenance Therapy With the Standard of Care (SoC) in Patients With Metastatic Non-Small Cell Lung Cancer (NSCLC), EGFR Wild Type
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SciClone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCI-Ta1-NSCLC-CHEMO P2-001
Record Dates: First submitted 2016-09-06; First posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: EGFR Wild Type; Thymosin Alpha 1; Non-Small Cell Lung Cancer; Thymalfasin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Thymalfasin; Trace amine-associated receptor 1; Drug Therapy; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thymalfasin (Thymosin alpha 1, Ta1) (Experimental): Arm A: 70 patients will receive Thymosin alpha 1 in 1mL SC injection five times a week (first four months); then two times a week for eight months. SoC chemotherapy and cisplatin (or carboplatin) for twelve months.
  Interventions: Drug: Thymalfasin (Thymosin alpha 1, Ta1); Drug: SoC (chemotherapy and platinum agent)
- SoC (chemotherapy and platinum agent) (Active Comparator): Arm B: 70 patients (control group) will receive SoC chemotherapy and cisplatin (or carboplatin) for twelve months.
  Interventions: Drug: SoC (chemotherapy and platinum agent)

INTERVENTIONS:
Drug: Thymalfasin (Thymosin alpha 1, Ta1) — Patients will be randomized to Thymosin alpha 1 plus SoC for treatment duration of 12 months. All patients will be followed for approximately 12 months or until the total number of PFS events required will be observed.
  Other Names: ZADAXIN
  Arms: Thymalfasin (Thymosin alpha 1, Ta1)
Drug: SoC (chemotherapy and platinum agent) — Patients will be randomized to SoC for treatment duration of 12 months. All patients will be followed for approximately 12 months or until the total number of PFS events required will be observed.
  Other Names: Pemetrexed, carboplatin or cisplatin

SUMMARY:
Thymosin alpha 1 plus maintenance therapy with the Standard of Care (SoC) chemotherapy plus cisplatin (or carboplatin) in patients with metastatic Non-Small Cell Lung Cancer (NSCLC), EGFR wild type

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histological or cytological confirmation of NSCLC (may be from initial diagnosis of NSCLC or subsequent biopsy). Only patients with available tissue samples may be included in the study (see major details in section 8 for the minimum sample characteristics)
* Activating mutations of EGFR diagnosis of Stage IIIB (with cytologically proven pleural effusion or pericardial effusion) or metastatic NSCLC, not amenable to curative surgery or radiotherapy
* Measurable disease by Response Evaluation Criteria in Solid Tumours (RECIST) in a lesion not previously irradiated or non-measurable disease (non measurable disease only for Phase I)
* Eastern Cooperative Oncology Group - performance status (ECOG-PS) 0-2
* Absolute neutrophil count (ANC) > 1.5 x 109/liter (L) and platelets > 100 x 109/L
* Bilirubin level either normal or <1.5 x ULN
* AST (SGOT) and ALT (SGPT) <2.5 x ULN (≤ 5 x ULN if liver metastases are present)
* Serum creatinine <1.5 x ULN
* Effective contraception for both, male and female patients, if the risk of conception exists
* Provision of written informed consent to the analysis of biological markers (registration)

Exclusion Criteria:

* Prior therapy with Thymosin alpha-1
* Prior chemotherapy for relapsed and/or metastatic NSCLC. Neoadjuvant/adjuvant chemotherapy is permitted if at least 12 months has elapsed between the end of chemotherapy and randomisation
* Prior treatment with Epidermal Growth Factor Receptor targeting small molecules or antibodies
* Radiotherapy within 14 days prior to drug administration, except as follows:
* Palliative radiation to organs other than chest may be allowed up to 2 weeks prior to drug administration, and
* Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling
* Patients with previously diagnosed and treated CNS metastases or spinal cord compression may be considered if they have evidence of clinically stable disease (SD) (no steroid therapy or steroid dose being tapered) for at least 28 days
* Patients with toxicities that have not come back (at least) to grade 1
* Pregnancy or suspected pregnancy
* Known severe hypersensitivity to TKI products
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* Any evidence of clinically active interstitial lung disease (ILD) (patients with chronic, stable, radiographic changes who are asymptomatic or patients with uncomplicated progressive lymphangitic carcinomatosis need not be excluded)
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
* As judged by the investigator, any inflammatory changes of the surface of the eye
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-05 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Time to progression free survival (PFS) | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (8):
  - Azienda Sanitaria Locale Frosinone, Frosinone
  - Istituto Nazionale dei Tumori, Milan
  - Roma_Campus Bio-Medico, Rome
  - Roma_Gemelli, Rome
  - Roma_Regina Apostolorum, Rome
  - Roma_Tor Vergata, Rome
  - Sant'Andrea Hospital, Rome
  - Presidio Sanitario San Camillo, Torino